CLINICAL TRIAL: NCT07145125
Title: Real-life Efficacy and Toxicity of Brentuximab-Vedotin Associated With Bendamustine in Patients With Relapsed or Refractory Hodgkin Lymphoma
Brief Title: Real-life Efficacy and Toxicity of Brentuximab-Vedotin Associated With Bendamustine in Patients With Relapsed or Refractory Hodgkin Lymphoma (HL-R2-B2)
Acronym: HL-R2-B2
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2024/60
Record Dates: First submitted 2025-03-18; First posted 2025-08-28 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2025-11

CONDITIONS: Relapsed or Refractory Hodgkin Lymphoma
Keywords: R/R Hodgkin lymphoma; Brentuximab-vedotin
MeSH Terms: conditions — Recurrence; Hodgkin Disease | interventions — Bendamustine Hydrochloride

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patient with relapsed or refractory Hodgkin Lymphoma
  Interventions: Drug: Brentuximab-Vedotin associated with Bendamustine

INTERVENTIONS:
Drug: Brentuximab-Vedotin associated with Bendamustine — Patient having received at least one course of the association Brentuximab-Vedotin and Bendamustine

SUMMARY:
Approximately 20% of patients diagnosed with Hodgkin lymphoma will eventually experience progression or relapse after first-line treatment, which carries a significant risk of disease-related death. Although several pilot studies have demonstrated high rates of sustained response with the combination of brentuximab vedotin (BV) and chemotherapy, consistent real-world data are still lacking. Moreover, there is no universally accepted salvage chemotherapy regimen in this setting, and clinical practices vary across centers. This study aims to describe the efficacy and toxicity of the BV + bendamustine (B2) regimen in patients with relapsed/refractory Hodgkin lymphoma (R/R HL) treated in France over a 10-year period, with or without an attempt at consolidative transplantation.

DETAILED DESCRIPTION:
This study is a retrospective observational multicentric study. All patients fulfilling inclusion criteria in participant centers will be included. Clinical data will be obtained from patients medical records.

ELIGIBILITY:
Inclusion Criteria:

* Patient with relapsed or refractory HL, after at least one first line of treatment
* Aged 18 years and over
* Having received at least one course of the Brenxutimab-Vedotin J1 and Bendamustine J1 + J2 combination

Exclusion Criteria:

* Minor patients
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with relapsed or refractory HL, after at least one first line of treatment
Sampling Method: Non-Probability Sample
Enrollment: 222 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-08-21 (Actual); Study Completion 2025-09-30 (Actual)

PRIMARY OUTCOMES:
Progression free survival (PFS) for the whole cohort | From date of inclusion until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 120 months
  Measured from the time of treatment initiation to the date of event : progression or death

SECONDARY OUTCOMES:
Overal survival (OS) for the whole cohort | From date of inclusion until the date of death from any cause assessed up to 120 months
  Measured from the time of treatment initiation to the date of death

CONTACTS AND LOCATIONS:
Locations (5):
- France (5):
  - CH de la Côte Basque, service Hématologie Clinique, Bayonne
  - CHU de Bordeaux, service Hématologie Clinique et Thérapie cellulaire, Bordeaux
  - CHU de Caen, service Hématologie Clinique, Caen
  - Institut Paoli Calmettes, service Hématologie Clinique, Marseille
  - CHU de Toulouse, service Hématologie Clinique, Toulouse

IPD SHARING:
Plan to Share IPD: No